CLINICAL TRIAL: NCT06487442
Title: Management of Postoperative Pain in France: a Prospective National Study
Acronym: ALGOSFAR2
Status: Completed | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: ALGOSFAR 2 / 2024-01
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Pain
Keywords: postoperative pain
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: No intervention, observation of postoperative pain scores and treatments

SUMMARY:
Managing postoperative pain is an ongoing challenge. Therefore, frequent surveys are needed to constantly evaluate and improve perioperative pain care. The French reference audit was published in 2008. Ten years later, the French AlgoSFAR survey of 70 centres and 3,315 patients highlighted a clear improvement in practices. However, these data have never been published in a referenced journal due to significant methodological biases.

In 2024, we do not have recent French data based on rigorous methodology in the field of postoperative pain management.

The objective of this study is to reassess postoperative pain management in France. This is a prospective national survey. The proposed methodology will make it possible to provide a relevant snapshot of the practices and quality of care. Secondarily, areas for improvement can be identified and these results will also help in the drafting of future recommendations.

100 centres representative of the French map of surgical centres will be contacted.

Inclusions will take place over 2 days, identical for all centres. All patients eligible for inclusion during this period will be included.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients benefiting of a scheduled surgery during the inclusion period in a participating centre.

Exclusion Criteria:

* Patients under 18 years old
* Patient's refusal
* Patients deprived of liberty
* Patients undergoing intracranial neurosurgery or cardiac surgery
* Expected surgery duration < 30 minutes
* urgent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for surgery
Sampling Method: Probability Sample
Enrollment: 3879 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Pain assessment | At rest over the first 3 days postoperatively
  Pain assessed with a numerical rating scale (NRS)

SECONDARY OUTCOMES:
Preoperative pain assessment | Preoperative assessment
  Pain assessed with a numerical rating scale (NRS)
Morphine consumption | Over the first 3 postoperative days
  Morphine consumption in mg
Frequency of administration of non-morphine analgesics | At rest over the first 3 days postoperatively
  Frequency of administration of non-morphine analgesics
Frequency of administration of regional anaesthesia | At rest over the first 3 days postoperatively
  Frequency of administration of regional anaesthesia
Frequency of postoperative nausea and vomiting (PONV) | At rest over the first 3 days postoperatively
  Frequency of postoperative nausea and vomiting (PONV)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Beloeil, MD, Principal Investigator — Société Française d'Anesthésie et de Réanimation
Locations (1):
- CHU Rennes - Hôpital Sud, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fletcher D, Fermanian C, Mardaye A, Aegerter P; Pain and regional anesthesia committee of the French Anesthesia and Intensive Care Society (SFAR). A patient-based national survey on postoperative pain management in France reveals significant achievements and persistent challenges. Pain. 2008 Jul 15;137(2):441-451. doi: 10.1016/j.pain.2008.02.026. Epub 2008 Apr 15. PMID 18417292
- [Result] Aubrun F, Langeron O, Quesnel C, Coriat P, Riou B. Relationships between measurement of pain using visual analog score and morphine requirements during postoperative intravenous morphine titration. Anesthesiology. 2003 Jun;98(6):1415-21. doi: 10.1097/00000542-200306000-00017. PMID 12766651
- [Result] Memtsoudis SG, Poeran J, Zubizarreta N, Cozowicz C, Morwald EE, Mariano ER, Mazumdar M. Association of Multimodal Pain Management Strategies with Perioperative Outcomes and Resource Utilization: A Population-based Study. Anesthesiology. 2018 May;128(5):891-902. doi: 10.1097/ALN.0000000000002132. PMID 29498951
- [Result] Beloeil H, Sion B, Rousseau C, Albaladejo P, Raux M, Aubrun F, Martinez V; SFAR research network. Early postoperative neuropathic pain assessed by the DN4 score predicts an increased risk of persistent postsurgical neuropathic pain. Eur J Anaesthesiol. 2017 Oct;34(10):652-657. doi: 10.1097/EJA.0000000000000634. PMID 28437260
- [Result] Fletcher D, Stamer UM, Pogatzki-Zahn E, Zaslansky R, Tanase NV, Perruchoud C, Kranke P, Komann M, Lehman T, Meissner W; euCPSP group for the Clinical Trial Network group of the European Society of Anaesthesiology. Chronic postsurgical pain in Europe: An observational study. Eur J Anaesthesiol. 2015 Oct;32(10):725-34. doi: 10.1097/EJA.0000000000000319. PMID 26241763
- [Result] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Result] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Result] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233